CLINICAL TRIAL: NCT05757804
Title: Study of 18F-0502B PET Imaging Targeting α-synuclein in the Diagnosis of α-synuclein-related Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, YiHui Guan, Professor, Huashan Hospital
Other Study IDs: KY2022-1065
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Positron-Emission Tomography; Alpha Synuclein Pathology
Keywords: Alpha Synuclein Pathology, Positron Emission Tomography
MeSH Terms: conditions — Synucleinopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-disease controls
- PD patients
- DLB patients
- MSA patients

SUMMARY:
To explore the diagnostic value of 18F-0502B brain imaging for α-Syn protein-related diseases in patients with PD. To evaluate the imaging range of α-Syn protein density in patients with α-Syn protein-related diseases and to assess the level of abnormal α-Syn protein deposition by PET imaging with this PET tracer, and its safety in human studies.

ELIGIBILITY:
Inclusion Criteria:

-

Non-disease controls:

1. Age between 60 and 80 years; gender is not limited.
2. Normal motor function as determined by the investigator through testing; UPDRS score of 0.
3. No neurological disease, major chronic disease, malignancy or acute infectious disease as confirmed by the investigator.
4. Informed consent must be signed in writing by the subject or his/her legal guardian or caregiver.
5. Blood count: white blood cell count (WBC) 4-10×109/L; platelets (PLT) 100-300×109/L; hemoglobin (HB) 120-160 g/L; renal function: serum creatinine less than or equal to the upper limit of the normal range; liver function: bilirubin, AST (SGOT)/ALT (SGPT) less than or equal to the upper limit of the normal range. Electrocardiogram: no significant abnormalities.
6. No neurological disorders, major chronic diseases, malignant tumors or acute infectious diseases as confirmed by the investigator, no family history of neurodegenerative movement disorders, no family history of neurological disorders related to movement disorders.
7. Be willing and able to cooperate with all the projects of this study.

PD patients:

1. Age between 60 and 80 years old; gender is not limited.
2. Patients meet the diagnostic criteria for PD (2015 version of the diagnostic guidelines for PD developed by the International Movement Disorders Society MDS), mild-moderate patients (H&Y classification 1-3 inclusive).
3. Brain MRI supports the diagnosis of PD and there is no other evidence of neurological disease.
4. No neurological disease, major chronic disease, malignancy or acute infectious disease as confirmed by the investigator.
5. Informed consent must be signed in writing by the subject or his/her legal guardian or caregiver.
6. Blood count: white blood cell count (WBC) 4-10×109/L; platelets (PLT) 100-300×109/L; hemoglobin (HB) 120-160 g/L; renal function: serum creatinine less than or equal to the upper limit of the normal range; liver function: bilirubin, AST (SGOT)/ALT (SGPT) less than or equal to the upper limit of the normal range. Electrocardiogram: no significant abnormalities.
7. No neurological disorders, major chronic diseases, malignant tumors or acute infectious diseases as confirmed by the investigator, no family history of neurodegenerative movement disorders, no family history of neurological disorders related to movement disorders.
8. Be willing and able to cooperate with all the projects of this study.

DLB patients:

1. Age was between 60 and 80 years; gender was not restricted.
2. Patients meet the diagnostic criteria for probable and likely Lewy body dementia developed by the International Working Group on Dementia with Lewy Bodies meeting
3. The diagnosis of DLB was supported by brain MRI and there was no other evidence of neurological disease.
4. No neurological disease, major chronic illness, malignancy, or acute infectious disease as confirmed by the investigator.
5. Informed consent must be signed in writing by the subject or his/her legal guardian or caregiver.
6. Blood count: white blood cell count (WBC) 4-10×109/L; platelets (PLT) 100-300×109/L; hemoglobin (HB) 120-160 g/L; renal function: serum creatinine less than or equal to the upper limit of the normal range; liver function: bilirubin, AST (SGOT)/ALT (SGPT) less than or equal to the upper limit of the normal range. Electrocardiogram: no significant abnormalities.
7. No neurological disorders, major chronic diseases, malignant tumors or acute infectious diseases as confirmed by the investigator, no family history of neurodegenerative movement disorders, no family history of neurological disorders related to movement disorders.
8. Be willing and able to cooperate with all the projects of this study.

MSA patients:

1. Age was between 60 and 80 years old; gender was not limited.
2. Patients meet the diagnostic criteria of the newly released 2022 MSA diagnostic consensus
3. Brain MRI supported the diagnosis of MSA and no other evidence of neurological disease.
4. No neurological disease, major chronic disease, malignancy, or acute infectious disease as confirmed by the investigator
5. Informed consent must be signed in writing by the subject or his/her legal guardian or caregiver.
6. Blood count: white blood cell count (WBC) 4-10×109/L; platelets (PLT) 100-300×109/L; hemoglobin (HB) 120-160 g/L; renal function: serum creatinine less than or equal to the upper limit of the normal range; liver function: bilirubin, AST (SGOT)/ALT (SGPT) less than or equal to the upper limit of the normal range. Electrocardiogram: no significant abnormalities.
7. No neurological disorders, major chronic diseases, malignant tumors or acute infectious diseases as confirmed by the investigator, no family history of neurodegenerative movement disorders, no family history of neurological disorders related to movement disorders.
8. Be willing and able to cooperate with all the projects of this study.

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from the study:

  1. Suffering from other serious neurological diseases, or gastrointestinal, cardiovascular, liver, kidney, blood system, tumor endocrine, respiratory system, immune deficiency and other serious diseases.
  2. In the past year, in addition to participating in the expected radiation exposure of this clinical study, have participated in other research programs or clinical care, resulting in radiation exposure exceeding the effective dose of 50 mSv.
  3. Liver function: bilirubin, AST(SGOT)/ALT(SGPT) less than or equal to the upper limit of the normal range.
  4. The candidate subject has received major surgery or received experimental drug or device treatment (with unclear effect or safety) within 1 month

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects were included from the neurology outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03-17 (Estimated); Primary Completion 2023-07-15 (Estimated); Study Completion 2024-01-14 (Estimated)

PRIMARY OUTCOMES:
Complete PET imaging | 90mins from time of injection
  Assessment of PET/CT imaging to detect α-synuclein in patients with α-synuclein-related Diseases

CONTACTS AND LOCATIONS:
Overall Officials: Fang Xie, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China